CLINICAL TRIAL: NCT01730118
Title: A Phase I Study of an Adenoviral Transduced Autologous Dendritic Cell Vaccine Expressing Human HER2/Neu ECTM in Adults With Tumors With 1-3+ HER2/Neu Expression
Brief Title: Ad/HER2/Neu Dendritic Cell Cancer Vaccine Testing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoyoung M. Maeng, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 130016; 13-C-0016
Record Dates: First submitted 2012-11-17; First posted 2012-11-21 (Estimated); Results first posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Breast Neoplasms; Breast Cancer; Adenocarcinomas; Metastatic Solid Tumors Characterized by HER2/Neu Expression
Keywords: Metastatic Solid Tumors; Human Epidermal Growth Factor Receptor 2 Expression (HER2/neu); Trastuzumab Exposure; Dendritic Cell Vaccine; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Adenocarcinoma | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 1/Part I dose escalation (Experimental): Adenoviral Transduced Autologous Human epidermal growth factor receptor (AdHER) dendritic cell (DC) vaccine administered at escalating doses
  Interventions: Biological: Adenoviral Transduced Autologous Human Epidermal Growth Factor Receptor (AdHER)2/neu Dendritic Cell (DC) Vaccine
- 2/Part I dose expansion (Experimental): Adenoviral Transduced Autologous Human epidermal growth factor receptor (AdHER) dendritic cell (DC) vaccine administered at a next lower dose or the highest dose
  Interventions: Biological: Adenoviral Transduced Autologous Human Epidermal Growth Factor Receptor (AdHER)2/neu Dendritic Cell (DC) Vaccine
- 3/Part 1 dose escalation (Experimental): Adenoviral Transduced Autologous Human epidermal growth factor receptor (AdHER) dendritic cell (DC) vaccine administered at Dose Level 1
  Interventions: Biological: Adenoviral Transduced Autologous Human Epidermal Growth Factor Receptor (AdHER)2/neu Dendritic Cell (DC) Vaccine
- 4/Part II dose escalation (Experimental): Adenoviral Transduced Autologous Human epidermal growth factor receptor (AdHER) dendritic cell (DC) vaccine administered at Dose Level 1
  Interventions: Biological: Adenoviral Transduced Autologous Human Epidermal Growth Factor Receptor (AdHER)2/neu Dendritic Cell (DC) Vaccine
- 5/Part II dose expansion (Experimental): Adenoviral Transduced Autologous Human epidermal growth factor receptor (AdHER) dendritic cell (DC) vaccine administered at Arm 1 maximum tolerated dose (MTD)
  Interventions: Biological: Adenoviral Transduced Autologous Human Epidermal Growth Factor Receptor (AdHER)2/neu Dendritic Cell (DC) Vaccine

INTERVENTIONS:
Biological: Adenoviral Transduced Autologous Human Epidermal Growth Factor Receptor (AdHER)2/neu Dendritic Cell (DC) Vaccine — autologous AdHER2 transduced dendritic cell vaccine manufactured under Good Manufacturing Practices (GMP) conditions from cryopreserved patient monocytes here at the National Institutes of Health (NIH) Clinical Center (CC) Department of Transfusion Medicine (DTM). Vaccine is administered intradermally at assigned dose level at weeks 0, 4, 8, 16 and 24 of the study.

SUMMARY:
Background:

- Human epidermal growth factor receptor 2 (HER2, also known as c-erbB2 or neu)/neu (HER2) is a tumor protein that appears in almost a third of breast cancers and in several other types of cancers such as colon, prostate and non-small cell lung. Tumors that overexpress HER2 can be associated with a more aggressive cancer, higher recurrence rates, and reduced survival rates. Researchers are testing a therapeutic cancer vaccine designed to stimulate the immune system to recognize HER2. The vaccine, called adenoviral transduced autologous human epidermal growth factor receptor (AdHER)/neu dendritic cell vaccine, is custom-made using an individual's own immune cells. These cells will be collected and used to produce the vaccine.

Objectives:

- To test the safety and effectiveness of AdHER2 vaccination.

Eligibility:

- Individuals at least 18 years of age who have HER2-expressing tumors.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies will also be performed.
* Participants will have an apheresis procedure to collect immune cells to create the vaccine.
* Participants will receive five doses of the vaccine at study Weeks 0, 4, 8, 16 and 24.
* Participants will be monitored with physical exams, frequent blood tests and imaging studies.

DETAILED DESCRIPTION:
Background:

* Human epidermal growth factor receptor 2 (HER2, also known as c-erbB2 or neu) is a proto-oncogene that encodes a 185-kd transmembrane tyrosine kinase receptor that participates in receptor-receptor interactions that regulate cell growth, differentiation and proliferation. Its over-expression contributes to neoplastic transformation.
* HER2 is over-expressed in up to 25-30% of node-positive or node-negative primary breast cancers and is associated with clinically aggressive breast cancer, a high recurrence rate and reduced survival.
* Trastuzumab (Herceptin (Registered trademark)) is a recombinant humanized mouse monoclonal antibody (MAb) that binds to the extracellular (EC) domain of the HER2 receptor. Its clinical efficacy is limited to patients with 3+ HER2 tumor expression documented by immunohistochemistry (IHC) or a Vysis fluorescent in situ hybridization (FISH) ratio of greater than 2.2. IHC is a subjective measurement of HER2/neu protein while FISH is an objective measurement of amplification of the HER2 oncogene.
* Although the use of trastuzumab has been associated with improved clinical outcomes, a significant number of patients are unresponsive to therapy and most eventually experience clinical progression. At present no vaccine is available that induces patients to make their own anti-HER2 antibodies.
* We propose to investigate the use of an adenoviral vector (Ad5f35) expressing human HER2ECTM (Ad5f35HER2ECTM- AdHER2) to transduce autologous dendritic cells for therapeutic vaccination in patients with HER2 expressing solid tumors.

Objectives:

-To determine the safety and toxicity of autologous AdHER2 dendritic cell vaccination.

Specifically, to determine if the fraction of patients with cancer therapeutics-related cardiac dysfunction (CTRCD), defined as a decrease in left ventricular ejection fraction (LVEF) >=10 percentage points, to a value LVEF to less than or equal to 53% (normal reference value for two-dimensional (2-D) echocardiography), is sufficiently low to warrant further development in subsequent trials.

-To determine the immunogenicity of autologous AdHER2 dendritic cell vaccination as measured by a 3-fold increase in anti-HER2/neu antibody concentration or a 4-fold increase in antibody dilution titers over baseline.

Study Design:

Open label, non-randomized, two-part, phase I study of 48 weeks duration for evaluation of primary endpoints with extended follow-up out to 30 months to monitor LVEF cardiac function.

Part I involves vaccine dose escalation in a population with no prior exposure to trastuzumab or other HER2-targeted therapies to determine if there is a significant, adverse safety signal regarding cardiac toxicity, in addition to preliminary assessment of the vaccine s immunogenicity and clinical activity. Five doses of 5, 10, 20 or 40 x 10(6) viable cells/AdHER2 DC vaccine will be given intradermally at Weeks 0, 4, 8, 16 and 24 in patients with metastatic solid tumors or high risk bladder cancer in the adjuvant setting Response will be evaluated by a Modified Immune- Related Response Criteria (irRC) based on Response Evaluation Criteria in Solid Tumors

(Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (modified irRC) at Weeks 8, 16, 24, 36 and 48 with confirmatory scans obtained not less than 4 weeks following initial documentation of objective response. Adjuvant bladder cancer patients will undergo re-staging at Weeks 8, 16, 24, 36 and 48 with confirmatory scans obtained not less than 4 weeks following initial documentation of objective response.

Part II is identical to part I, in the schedule of treatment and response evaluation, but is conducted in a population with prior exposure to trastuzumab and other HER2-targeted therapies.

Eligibility:

Part I:

* Adults >= 18 with recurrent, metastatic solid tumors for whom trastuzumab is not clinically indicated in standard of care OR who are naive to HER2 targeted therapies:
* Patients with ovarian, cervical, colon, non-small cell lung, renal cell, bladder and prostate cancer, and malignant soft tissue and bone tumor or other solid tumors that is HER2 1+, 2+ or 3+ by IHC OR have a Vysis FISH result greater than or equal to 1.8.

  * Patients with breast cancer that is HER2 1+ or 2+ by IHC or with a Vysis FISH result less than or equal to 1.8 - less than or equal to 2.2.
  * Measurable disease, with the exception of metastatic bladder cancer patients that have completed first line chemotherapy and may not have measurable disease.
* Adults greater than or equal to 18 with HER2+ bladder cancer in the adjuvant setting

  * Tumor stage T3a, T3b, T4a and T4b or any node positive disease.
  * Tumors that are HER2 1+, 2+ or 3+ by IHC or have a Vysis FISH result greater than or equal to 1.8.
  * greater than or equal to 6 weeks status post primary surgery with curative intent.
  * Eastern Cooperative Oncology Group (ECOG) 0-1.
  * Naive to trastuzumab, pertuzumab, lapatinib, ado-trastuzumab emtansine (TDM1) or other HER2-directed therapies.

Part II:

* Adults >= 18 with breast, gastric or gastroesophageal junction or other cancers with 1+ to 3+ HER2/neu expression by IHC or a Vysis FISH result > 2.2.
* Recurrent metastatic disease, ECOG 0-1. Disease progression following HER2-targeted therapies. i.e., trastuzumab, pertuzumab, lapatinib, ado-trastuzumab emtansine or other HER2 agents.
* Measurable disease.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Common Eligibility for Parts I and II

* Adults greater than or equal to 18 with malignant soft tissue and bone tumors and recurrent or progressive, metastatic solid tumors who have progressed on standard therapies except in adjuvant for high risk bladder cancer in Part I.
* Recurrent or progressive disease on prior standard therapies with known clinical benefit with the exception of adjuvant bladder cancer population.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-1.
* Baseline left ventricular ejection fraction (LVEF) by two-dimensional (2D) Echocardiogram greater than or equal to 53%.
* Greater than or equal to 1 week since standard or investigational treatment for metastatic disease.
* Stable, concurrent use of hormone therapy for hormone receptor positive breast cancer is permitted.
* Hematologic parameters: absolute neutrophil count (ANC) greater than or equal to 1000 cells/mm^3, absolute lymphocyte count (ALC) greater than or equal to 300 cells/mm^3, Hemoglobin greater than or equal to 9.0 gm/dL, white blood cell (WBC) greater than or equal to 2,500 cells/mm^3, platelet count greater than or equal to 75,000/mm^3, prothrombin time (PT)/partial thromboplastin time (PTT) less than or equal to 1.5X the upper limits of normal.
* Chemistry parameters: Creatinine less than or equal to 1.5 mg/dL, serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) less than or equal to 3X the upper limits of normal and total bilirubin less than or equal to 1.5 mg/dl, Alkaline phosphatase (Alk PO4) less than or equal to 3X the upper limits of normal (except for patients with documented metastatic disease to bone and/or liver).
* Negative serum beta human chorionic gonadotropin (HCG) if female and of childbearing potential.
* Negative human immunodeficiency virus (HIV) 1/2 serology and sample drawn for human T-cell lymphotropic virus (HTLV). Patients with HIV are excluded from participating on this clinical trial because their immunodeficiency would confound the evaluation of adverse events which would hinder meeting the primary objective.
* Negative serology for hepatitis B and C unless the result is consistent with prior vaccination or prior infection with full recovery.
* Willingness of female and male subjects to use effective contraception e.g., oral contraceptives, barrier device, intrauterine device, or condoms, during the study and for three months following the last dose of study vaccine. We suggest that subjects do not become pregnant or father a child during the study, and for 3 months following receipt of the investigational adenoviral transduced autologous human epidermal growth factor receptor (AdHER) dendritic cell (DC) vaccine.
* Able to understand and provide Informed Consent.
* Patients with 1+ to 3+ human epidermal growth factor receptor 2 (HER2)/neu expression by immunohistochemistry (IHC) or an equivocal or positive fluorescence in situ hybridization (FISH) result by 2013 American Society of Clinical Oncology (ASCO)/Corrective Action Plan (CAP) guideline.
* Patients must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

Part I Eligibility

* Naive to trastuzumab (Herceptin), pertuzumab (Perjeta) and lapatinib (Tykerb), ado-trastuzumab emtansine (Kadcyla) or other HER2-directed therapies.
* Malignancy as follows:
* Malignant soft tissue and bone tumors and recurrent or progressive, metastatic solid tumors who have progressed on standard therapies; or,
* Bladder cancer in the adjuvant setting (adjuvant bladder cancer patients):

  * Tumor stage T3a, T3b, T4a, T4b and any node positive disease regardless of tumor stage.
  * Status-post primary cystectomy with curative intent.
  * May or may not have received neoadjuvant cisplatin-based combination chemotherapy per National Comprehensive Cancer Network (NCCN) guidelines.
  * May or may not have received adjuvant radiotherapy or chemotherapy based on pathologic risk per NCCN guidelines.
  * Greater than or equal to 6 weeks s/p primary surgery with curative intent.
* NOTE: Patients with breast, ovarian, cervical, colon, gastric/gastroesophageal junction, non-small cell lung, renal cell, bladder, malignant soft tissue and bone tumor, prostate cancer or other solid tumors.

Part II Eligibility

* Malignant soft tissue and bone tumors and recurrent or progressive, metastatic solid tumors who have progressed on standard therapies.
* Recurrent or progressive metastatic disease after standard of care HER2-targeted therapies, i.e., trastuzumab (Herceptin), pertuzumab (Perjeta), lapatinib (Tykerb), ado-trastuzumab emtansine (TDM1) (Kadcyla) or other HER2-directed therapies.
* Stable, concurrent use of tamoxifen or aromatase inhibitors for hormone receptor positive breast cancer is permitted.

EXCLUSION CRITERIA:

* Pregnant women are excluded from this study because Adenoviral Transduced Autologous Human epidermal growth factor receptor (AdHER) dendritic cell (DC) vaccine may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AdHER DC vaccine, breastfeeding should be discontinued if the mother is treated with AdHER DC vaccine.
* Patients with active central nervous system (CNS) metastases or leptomeningeal involvement by tumor (patients with a history of brain metastases who have successfully treated for brain metastasis by surgery or radiation and who have not had any evidence of the new or progressive CNS disease for more than 12 months are eligible).
* Patients with rapidly progressing disease in the opinion of the Principal Investigator.
* Patients with inadequate bilateral peripheral venous or central venous catheter access for the required apheresis to allow generation of the autologous AdHER2 DC vaccine product.
* Clinically significant cardiac dysfunction defined as a history of > New York Heart Association (NYHA) Class II symptoms, angina, congestive heart failure, myocardial infarction, arrhythmias or cardiac dysfunction requiring treatment or discontinuation of chemotherapy.
* History of changes in baseline LVEF that occurred during prior treatment with anti-HER2 treatment.
* Cumulative doxorubicin dose > 400mg/m^2 (>450 mg/m^2 for malignant soft tissue and bone tumor patients) or cumulative epirubicin dose > 800mg/m^2.
* Use of any standard chemotherapy or other investigational agent(s) within 1 week of study enrollment.
* Use of systemic corticosteroid therapy within 2 weeks of study enrollment, including patients receiving replacement corticosteroid therapy. Note: only topical, inhaled and intranasal steroid therapy is permitted.
* Active systemic viral, bacterial or fungal infection requiring treatment.
* A medical history which the treating physician believes causes the patient to be excluded. This includes a remote history of cancer. Please note: Squamous cell carcinoma, basal cell carcinoma and remote history of cancer with no evidence of recurrence for the past 5 years are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung M Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Moasser MM. The oncogene HER2: its signaling and transforming functions and its role in human cancer pathogenesis. Oncogene. 2007 Oct 4;26(45):6469-87. doi: 10.1038/sj.onc.1210477. Epub 2007 Apr 30. PMID 17471238
- [Background] Wolff AC, Hammond ME, Schwartz JN, Hagerty KL, Allred DC, Cote RJ, Dowsett M, Fitzgibbons PL, Hanna WM, Langer A, McShane LM, Paik S, Pegram MD, Perez EA, Press MF, Rhodes A, Sturgeon C, Taube SE, Tubbs R, Vance GH, van de Vijver M, Wheeler TM, Hayes DF; American Society of Clinical Oncology; College of American Pathologists. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for human epidermal growth factor receptor 2 testing in breast cancer. J Clin Oncol. 2007 Jan 1;25(1):118-45. doi: 10.1200/JCO.2006.09.2775. Epub 2006 Dec 11. PMID 17159189
- [Background] Lan KH, Lu CH, Yu D. Mechanisms of trastuzumab resistance and their clinical implications. Ann N Y Acad Sci. 2005 Nov;1059:70-5. doi: 10.1196/annals.1339.026. PMID 16382045
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0016.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs): Vaccine is administered intradermally at assigned dose level at weeks 0, 4, 8, 16, and 24 of study.
  5x10^6 Total Nucleated Cells (TNCs)
- Part I Dose Escalation Level 2 - 10x10^6 Total Nucleated Cells (TNCs): Vaccine is administered intradermally at assigned dose level at weeks 0, 4, 8, 16, and 24 of study.
  10x10^6 Total Nucleated Cells (TNCs)
- Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs); Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs): Vaccine is administered intradermally at assigned dose level at weeks 0, 4, 8, 16, and 24 of study.
  20x10^6 Total Nucleated Cells (TNCs)
- Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs); Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs): Vaccine is administered intradermally at assigned dose level at weeks 0, 4, 8, 16, and 24 of study.
  40x10^6 Total Nucleated Cells (TNCs)
- Enrolled But Not Treated: Participants were enrolled on the study but not treated.
Period: Dose Escalation
Arm/Group | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 2 - 10x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Enrolled But Not Treated
Started | 6 | 7 | 6 | 6 | 0 | 0 | 2
Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 6 | 7 | 3 | 6 | 0 | 0 | 2
Not completed — Death on study | 5 | 7 | 2 | 6 | 0 | 0 | 0
Not completed — Died before treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Chose to start a different treatment | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Disease progression prior to treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Dose Expansion
Arm/Group | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 2 - 10x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Enrolled But Not Treated
Started | 0 | 0 | 0 | 0 | 3 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 3 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other medical condition | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Inability to return | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 2 - 10x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Enrolled But Not Treated | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 3 | 3 | 2 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 3 | 3 | 3 | 3 | 1 | 25
  >=65 years | 1 | 0 | 3 | 3 | 0 | 0 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.28 (10.21) | 57.1 (7.92) | 64.5 (6.3) | 62.65 (5.08) | 60.03 (2.11) | 56.33 (7.62) | 63.9 (11.74) | 58.46 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 5 | 1 | 1 | 0 | 21
  Male | 2 | 1 | 2 | 1 | 2 | 2 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 7 | 6 | 6 | 3 | 3 | 2 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 6 | 5 | 6 | 5 | 3 | 2 | 1 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 6 | 6 | 3 | 3 | 2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiac Toxicity
Description: Cardiac toxicity defined as cardiac dysfunction due to damage to the heart muscles or valves. Cardiac toxicity was assessed by serial echocardiography to determine left ventricular ejection fraction (LVEF) at baseline and following receipt of the last dose of vaccine. Cardiac toxicity is at least a 10% decline from the baseline in cardiac function. Normal LVEF is >-53%. Below 53% is a cardiac dysfunction.
Time Frame: Baseline through receipt of last dose of vaccine, up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 2 - 10x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs)
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 3 | 3
Participants
  Normal LVEF >-53% | 6 | 7 | 6 | 6 | 3 | 3
  Cardiac Dysfunction - LVEF below 53% | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Develop at Least a 4-fold or 2.5- Fold Increase in Anti-Human Epidermal Growth Factor Receptor (HER2)/Neu Antibody Dilution Titers
Description: Vaccine immunogenicity was determined by the number of participants who develop at least a 4-fold increase in antibody dilution titers over baseline at the time points measured. The antibody response following the vaccination was assessed using peptide-array and reported as fold increase compared to the baseline values using the cut-off of 4 fold per study definition of the vaccine immunogenicity and also of 2.5 fold to aid the interpretation of the result.
Time Frame: Baseline through last dose of vaccine, up to 24 weeks
Population: Not all participants had samples for analyses. Samples from 13 participants were analyzed in the following groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 2 - 10x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs)
Number analyzed (Participants) | 1 | 4 | 4 | 4 | 0 | 0
Participants
  4-fold Increase | 0 | 0 | 1 | 0 | 0 | 0
  2.5- fold Increase | 0 | 1 | 2 | 1 | 0 | 0

3. Secondary Outcome: Number of Participants Who Experienced Tumor Shrinkage or Stabilization That is Sufficient by Modified Immune Response Related Criteria (irRC) to be Considered Stable Disease (SD), a Partial Response (PR) or Better (Complete Response (CR)
Description: Number of participants who experienced tumor shrinkage or stabilization that is sufficient by modified immune response related criteria (irRC) to be considered stable disease (SD), a partial response (PR) or better (complete response (CR). SD is neither partial response nor progressive disease (PD). PR is ≥ 30% decrease in tumor burden compared with baseline, confirmation required. CR is disappearance of all target and non-target lesions. Lymph nodes must regress to <10mm short axis. No new lesions, confirmation required. PD ≥ 20% increase in tumor burden compared with baseline, with nadir, or reset baseline. New lesions added to the tumor burden, confirmation required.
Time Frame: At 8, 16, 24, 36, 48, 76, 100, and 124 weeks after initial vaccination
Population: Not all participants were available for analyses. Twenty one participants were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 2 - 10x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs)
Number analyzed (Participants) | 5 | 7 | 3 | 4 | 1 | 1
Participants
  Stable Disease at Week 8 | 0 | 2 | 1 | 1 | 0 | 1
  Partial Response at Week 8 | 0 | 1 | 1 | 0 | 0 | 0
  Complete Response at Week 8 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease at Week 16 | 0 | 2 | 1 | 1 | 0 | 1
  Partial Response at Week 16 | 0 | 1 | 1 | 0 | 0 | 0
  Complete Response at Week 16 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease at Week 24 | 0 | 0 | 1 | 1 | 0 | 1
  Partial Response at Week 24 | 0 | 0 | 0 | 0 | 0 | 0
  Complete Response at Week 24 | 0 | 0 | 1 | 0 | 0 | 0
  Stable Disease at Week 36 | 0 | 0 | 1 | 0 | 0 | 0
  Partial Response at Week 36 | 0 | 0 | 0 | 0 | 0 | 0
  Complete Response at Week 36 | 0 | 0 | 1 | 0 | 0 | 0
  Stable Disease at Week 48 | 0 | 0 | 1 | 0 | 0 | 0
  Partial Response at Week 48 | 0 | 0 | 0 | 0 | 0 | 0
  Complete Response at Week 48 | 0 | 0 | 1 | 0 | 0 | 0
  Stable Disease at Week 76 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response at Week 76 | 0 | 0 | 0 | 0 | 0 | 0
  Complete Response at Week 76 | 0 | 0 | 1 | 0 | 0 | 0
  Stable Disease at Week 100 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response at Week 100 | 0 | 0 | 0 | 0 | 0 | 0
  Complete Response at Week 100 | 0 | 0 | 1 | 0 | 0 | 0
  Stable Disease at Week 124 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response at Week 124 | 0 | 0 | 0 | 0 | 0 | 0
  Complete Response at Week 124 | 0 | 0 | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 29 months and 13 days, 28 months and 28 days, 40 months and 2 days, 24 months and 23 days, 25 months and 30 days, and 28 months and 3 days for each group respectively.
Measure: Count of Participants; unit: Participants
Groups:
- Part I Dose Escalation Level 3 - 520x10^6 Total Nucleated Cells (TNCs); Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs): Vaccine is administered intradermally at assigned dose level at weeks 0, 4, 8, 16, and 24 of study.
  20x10^6 Total Nucleated Cells (TNCs)
Arm/Group | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 2 - 10x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 3 - 520x10^6 Total Nucleated Cells (TNCs) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Enrolled But Not Treated
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 3 | 3 | 2
Participants | 6 | 7 | 6 | 6 | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 29 months and 13 days, 28 months and 28 days, 40 months and 2 days, 24 months and 23 days, 25 months and 30 days, and 28 months and 3 days for each group respectively.
Groups:
- Part I Dose Escalation Level 2 -10x10^6 Total Nucleated Cells (TNCs): Vaccine is administered intradermally at assigned dose level at weeks 0, 4, 8, 16, and 24 of study.
  10x10^6 Total Nucleated Cells (TNCs)
Arm/Group | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 2 -10x10^6 Total Nucleated Cells (TNCs) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) | Enrolled But Not Treated
All-Cause Mortality (participants affected / at risk) | 5/6 | 7/7 | 2/6 | 6/6 | 1/3 | 0/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 5/6 | 7/7 | 2/6 | 6/6 | 1/3 | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 6/6 | 6/6 | 2/3 | 3/3 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) (N=6) | Part I Dose Escalation Level 2 -10x10^6 Total Nucleated Cells (TNCs) (N=7) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) (N=6) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) (N=6) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) (N=3) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) (N=3) | Enrolled But Not Treated (N=2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (6) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 5 (5) | 7 (7) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (16) | 0 (0) | 1 (2) | 0 (0)
Fever (General disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (48) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (18) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, left renal abscess (Infections and infestations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (10) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I Dose Escalation Level 1 - 5x10^6 Total Nucleated Cells (TNCs) (N=6) | Part I Dose Escalation Level 2 -10x10^6 Total Nucleated Cells (TNCs) (N=7) | Part I Dose Escalation Level 3 - 20x10^6 Total Nucleated Cells (TNCs) (N=6) | Part II Dose Escalation Level 1 - 20x10^6 Total Nucleated Cells (TNCs) (N=6) | Part I Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) (N=3) | Part II Dose Expansion Cohort - 40x10^6 Total Nucleated Cells (TNCs) (N=3) | Enrolled But Not Treated (N=2)
Abdominal distension (Gastrointestinal disorders) | 1 (5) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 3 (12) | 4 (47) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (5) | 1 (14) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (8) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (10) | 3 (30) | 1 (4) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (30) | 2 (27) | 2 (30) | 2 (36) | 1 (5) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (21) | 0 (0) | 3 (32) | 2 (15) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (12) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 2 (15) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (15) | 2 (11) | 1 (4) | 1 (35) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (11) | 1 (24) | 1 (6) | 1 (12) | 1 (20) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (7) | 1 (6) | 1 (15) | 0 (0) | 1 (10) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, Swollen lymph nodes. Left supraclavical area. (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (5) | 1 (4) | 1 (25) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (21) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 2 (45) | 0 (0) | 0 (0) | 1 (13) | 0 (0)
Cardiac disorders - Other, Mid RV dilation (Cardiac disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (12) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (9) | 2 (9) | 1 (30) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (6) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 1 (20) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (13) | 3 (14) | 1 (4) | 2 (44) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (5) | 2 (10) | 1 (15) | 0 (0) | 1 (15) | 1 (13) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (5) | 2 (10) | 0 (0) | 1 (12) | 1 (5) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (10) | 1 (15) | 1 (12) | 2 (15) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (9) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 2 (18) | 1 (4) | 4 (54) | 0 (0) | 1 (2) | 0 (0)
Edema limbs (General disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (8) | 1 (5) | 0 (0) | 0 (0)
Eye disorders - Other, Look like fleas/consult ophthalmology (Eye disorders) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, Transient light flashes in eyes (Eye disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, Specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Transient visual field defect L eye associated with flashes, lasting < 2 minutes.
Fatigue (General disorders) | 3 (13) | 4 (47) | 3 (23) | 6 (61) | 1 (10) | 1 (2) | 0 (0)
Fever (General disorders) | 2 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (10) | 0 (0) | 1 (15) | 1 (24) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 1 (13) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (5) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Epigastric abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Left sided abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (5) | 1 (7) | 2 (41) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (10) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (20) | 1 (6) | 1 (4) | 1 (5) | 1 (10) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (10) | 1 (6) | 3 (62) | 4 (57) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Cyst R-scapular (Infections and infestations) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Pneumocystis carina pneumonia or PJP (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 5 (85) | 7 (277) | 5 (513) | 6 (396) | 2 (70) | 3 (138) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (15) | 2 (24) | 1 (5) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (20) | 0 (0) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (20) | 2 (34) | 4 (189) | 4 (42) | 2 (15) | 1 (13) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (12) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (24) | 0 (0) | 1 (26) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (13) | 3 (18) | 1 (13) | 2 (36) | 1 (5) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 1 (10) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 1 (13) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (13) | 2 (41) | 3 (88) | 2 (10) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (5) | 1 (12) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (15) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (14) | 0 (0) | 0 (0) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Renal and urinary disorders - Other, Ciprofloxacine 250mg twice a day for 5 days (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0)
Renal and urinary disorders - Other, Pyruria on Levaquin (Renal and urinary disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Serum amylase increased (Infections and infestations) | 0 (0) | 1 (12) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Itching around ears bilateral- Dr. Bronner's Magic Soaps
Skin and subcutaneous tissue disorders - Other, Left inguinal itch and redness. (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0) — Skin coloration change-Right arm. Patient reported noticing the change after 1st vaccine.
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, right nephrostomy placement, ureteroscopy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (42) | 1 (30) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (19) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (38) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (5) | 5 (24) | 1 (13) | 1 (12) | 1 (5) | 1 (2) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (5) | 4 (21) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (4) | 0 (0) | 2 (30) | 0 (0) | 1 (10) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT01730118/Prot_SAP_000.pdf
  • Informed Consent Form: Standard Consent (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT01730118/ICF_001.pdf
  • Informed Consent Form: Addendum to 13C0016 Consent (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT01730118/ICF_002.pdf